CLINICAL TRIAL: NCT07023302
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Efficacy and Safety of Upadacitinib in Adult and Adolescent Subjects With Alopecia Areata and at Least 25% Scalp Hair Loss
Brief Title: A Study to Evaluate the Safety and Effectiveness of Upadacitinib Tablets in Adult and Adolescent Participants in Japan With Alopecia Areata
Acronym: Jump Up AA JP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M24-600
Record Dates: First submitted 2025-06-10; First posted 2025-06-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Upadacitinib; JUMP-UP; AA
MeSH Terms: conditions — Alopecia Areata | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Group 1A: Upadacitinib Dose A (Experimental): Participants will receive upadacitinib dose A once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Group 2A: Upadacitinib Dose B (Experimental): Participants will receive upadacitinib dose B once daily for 52 weeks in Period A and Period B.
  Interventions: Drug: Upadacitinib
- Group 3A: Upadacitinib Placebo (Placebo Comparator): Participants will receive upadacitinib placebo once daily for 24 weeks in Period A.
  Interventions: Drug: Upadacitinib Placebo
- Group 1B: Upadacitinib Dose A (Experimental): Participants initially randomized to placebo (Period A) will be re-randomized to receive upadacitinib dose A once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Group 2B: Upadacitinib Dose B (Experimental): Participants initially randomized to placebo (Period A) will be re-randomized to receive upadacitinib dose B once daily for 28 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Period C: Upadacitinib Dose A Remains Dose A (Experimental): For participants initially randomized to dose A in Periods A and B and participants initially randomized to placebo who switched to dose A in Period B: participants with a Severity of Alopecia Tool (SALT) score <= 10 at Week 52 (end of Period B) will remain on blinded upadacitinib dose A once daily in Period C for 52 weeks.
  Interventions: Drug: Upadacitinib
- Period C: Upadacitinib Dose A to Dose B (Experimental): For participants initially randomized to dose A in Periods A and B and participants initially randomized to placebo who switched to dose A in Period B: participants with a SALT score > 10 at Week 52 (end of Period B) will dose escalate to blinded upadacitinib dose B once daily in Period C for 52 weeks.
  Interventions: Drug: Upadacitinib
- Period C: Upadacitinib Dose B Non-Sustained Responders (Experimental): For participants initially randomized to dose B in Periods A and B and participants initially randomized to placebo who switched to dose B in Period B: participants with a SALT score > 10 at Week 40 or Week 52 will remain on blinded upadacitinib dose B once daily in Period C for 52 weeks.
  Interventions: Drug: Upadacitinib
- Period C: Upadacitinib Dose B Sustained Responders (Experimental): For participants initially randomized to dose B in Periods A and B and participants initially randomized to placebo who switched to dose B in Period B: participants with a SALT score <= 10 at Week 40 and Week 52 will receive blinded upadacitinib dose A once daily in Period C for 52 weeks.
  Interventions: Drug: Upadacitinib
- Period C: Open-Label Upadacitinib Dose B (Experimental): Participants with no improvement or worsening from Baseline in their SALT score at the Week 40 visit or any scheduled visit thereafter will receive open-label upadacitinib dose B once daily for 52 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Arms: Group 1A: Upadacitinib Dose A; Group 1B: Upadacitinib Dose A; Group 2A: Upadacitinib Dose B; Group 2B: Upadacitinib Dose B; Period C: Open-Label Upadacitinib Dose B; Period C: Upadacitinib Dose A Remains Dose A; Period C: Upadacitinib Dose A to Dose B; Period C: Upadacitinib Dose B Non-Sustained Responders; Period C: Upadacitinib Dose B Sustained Responders
Drug: Upadacitinib Placebo — Oral Tablets
  Arms: Group 3A: Upadacitinib Placebo

SUMMARY:
Alopecia areata (AA) is a disease that happens when the immune system attacks hair follicles and causes hair loss. AA usually affects the head and face, but hair loss can happen on any part of the body. The purpose of this study is to assess how safe, effective, and tolerable upadacitinib is in adolescent and adult participants in Japan with severe AA.

Upadacitinib is an approved drug being investigated for the treatment of AA. In Period A, participants are placed in 1 of 3 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to placebo. In Period B, participants originally randomized to a upadacitinib dose group in Period A will continue their same treatment in Period B. Participants originally randomized to Placebo in Period A will be re-randomized in 1 of 2 groups receiving upadacitinib. Participants who complete Period B can join Period C and will receive 1 of 2 doses of upadacitinib for up to 52 weeks based on their SALT score. Around 123 adolescent and adult participants with severe AA will be enrolled in the study at approximately 20 sites in Japan.

Participants will receive oral tablets of either upadacitinib or placebo once daily for up to 104 weeks with the potential of being re-randomized into a different treatment group at Weeks 24 and 52. Participants will be followed up for up to 30 days after their last study drug dose.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health as determined by the Principal Investigator, based upon the results of the Screening assessments and medical history.
* Diagnosis of severe alopecia areata (AA) with Severity of Alopecia Tool (SALT) score >= 25 (>= 25% scalp hair loss) at Screening and Baseline.
* Current episode of AA of less than 8 years.

Exclusion Criteria:

* Current diagnosis of primarily diffuse type of AA.
* Current diagnosis of other types of alopecia that would interfere with evaluation of AA, including but not limited to female pattern hair loss, male pattern hair loss (androgenetic alopecia) Stage III or greater based on Hamilton-Norwood classification, traction alopecia, lichen planopilaris (LPP), discoid lupus, frontal fibrosing alopecia (FFA), central centrifugal cicatricial alopecia (CCCA), folliculitis decalvans, trichotillomania, and telogen effluvium.
* Diagnosis of other types of inflammatory scalp, eyebrow, or eyelash disorders that would interfere with evaluation of AA as determined by the investigator, including but not limited to seborrheic dermatitis, scalp psoriasis, atopic dermatitis (AD), and tinea capitis.
* Active infection(s) requiring treatment with intravenous anti-infectives within 30 days, or oral/intramuscular anti-infectives within 14 days prior to the Baseline Visit.
* Chronic recurring infection and/or active viral infection that, based on the investigator's clinical assessment, makes the participant an unsuitable candidate for the study.

Ages: 12 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with the Achievement of Severity of Alopecia Tool (SALT) Score <= 10 | Week 24
  The SALT is a global alopecia areata (AA) severity score based on the combination of extent and density of scalp hair loss. The score is determined by visually defining the amount of terminal hair loss in each of the 4 views of the scalp (left and right side each accounting for 18% of scalp area, the top for 40%, and the back for 24%) and adding these together with a maximum score of 100%. A SALT score of <= 10 is defined as less than or equal to 10% hair loss.
Number of Participants with Adverse Events (AEs) | Up to approximately 108 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants with the Achievement of Patient-Reported Outcome (PRO) for Scalp Hair Assessment of 0 or 1 | Week 24
  The PRO for Scalp Hair Assessment is single item, five-point, categorical response scale that asks respondents to look in the mirror and assess the total area of the scalp with missing hair. Response items range from "No missing hair" to "Nearly all or all" and includes percentage ranges for each category (0%, 1 to 20%, 21 to 49%, 50 to 94%, and 95 to 100%). Responses among participants with baseline score >=2.
Percentage of Participants with the Achievement of Patients' Global Impression of Change of Alopecia Areata (PaGIC-AA) Score of 1 "Much Better" or 2 "Moderately Better" | Week 24
  The PaGIC-AA is a single-item measure that asks participants to rate how their alopecia condition has changed overall since the start of the study using a 7-point scale. Responses range from "much better" to "much worse."

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- Japan (15):
  - Nagoya City University Hospital /ID# 275409, Nagoya, Aichi-ken
  - Kurume University Hospital /ID# 275519, Kurume-shi, Fukuoka
  - Kanazawa Medical University Hospital /ID# 275521, Kahoku-gun, Ishikawa-ken
  - Nagomi Dermatology Clinic /ID# 275418, Ebina-shi, Kanagawa
  - Rifu Dermatology Allergy Clinic /ID# 274875, Miyagi-gun, Miyagi
  - Tohoku University Hospital /ID# 274931, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 274775, Niigata, Niigata
  - Shinsaibashi Inui Dermatology Clinic /ID# 274851, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 274956, Osaka, Osaka
  - Hamamatsu University Hospital /ID# 274639, Hamamatsu, Shizuoka
  - Kyorin University Hospital /ID# 274882, Mitaka-shi, Tokyo
  - Tokyo Medical University Hospital /ID# 274844, Shinjuku-ku, Tokyo
  - Keio University Hospital /ID# 275640, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital /ID# 274638, Ube, Yamaguchi
  - Juntendo Tokyo Koto Geriatric Medical Center /ID# 275424, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-600